CLINICAL TRIAL: NCT04861753
Title: The Effects of Reiki and Back Massage on the Pain and Vital Signs of Women After Abdominal Hysterectomy: A Randomized Controlled Trial
Brief Title: The Effects of Reiki and Back Massage on the Pain and Vital Signs
Status: Completed | Type: Observational
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, HEDİYE UTLİ, PhD, RN, Assistant Professor, Mardin Artuklu University
Other Study IDs: ArtukluU
Record Dates: First submitted 2021-04-05; First posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pain; Abdominal Pain
Keywords: Back massage; Hysterectomy; Pain; Reiki
MeSH Terms: conditions — Pain; Abdominal Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Reiki: The modern-day Reiki (pronounced "ray-kee") practiced in the United States originated in Japan with Mikao Usui in the early 1900s. Reiki is a complementary and adjuvant therapeutic technique. Reiki, which is classified as an "energy healing therapy", is a technique of channeling universal energy in order to reduce stress, promote relaxation, and enhance well-being.
  Interventions: Other: Reiki and back massage
- Back massage: Massage therapy involves the manipulation of the soft tissues of the body by touch. It consists of gentle movements such as effleurage, petrissage and percussion.
  Interventions: Other: Reiki and back massage
- Control: Routine postoperative care was given to the control group without any intervention

INTERVENTIONS:
Other: Reiki and back massage — In the current study, at the beginning of the treatment, the researcher held his hands 2-3 cm above the patient sand adjusted the aura of the patient by making circular movements from the head to the feet. After this process of aura attunement, the researcher placed his hands directly on the patient's body. In the areas where the practitioner had placed his hands for an average of three minutes, starting from between the eyes, the researcher felt various degrees of warmth and tingling in his palms. Only the back was left exposed to prevent the patient becoming cold. The researcher took a little non-aromatic baby oil in hand and heated it, then began a 20-minute-long massage. The massage consisted of 6.5 minutes of effleurage (stroking), 3.5 minutes of petrissage (kneading), 13 minutes of effleurage and seven minutes of petrissage.
  Groups: Back massage; Reiki

SUMMARY:
The practice of Reiki and back massage applications in support of pharmacological treatment is among the nursing initiatives and these practices increase the autonomy of the profession. The aim of this study was to determine the effects of Reiki and back massage on pain, analgesic use and vital signs in women who had undergone open abdominal hysterectomy. This was an experimental study with a single, blinded, pretest-posttest control group. The population of the study consisted of women who had abdominal hysterectomy in the Obstetrics Clinics at Gazi Yasargil Training and Research Hospital and Dicle University Hospital between July 2017 and February 2018. The patients were divided into three groups: Reiki, back massage and control, with 34 patients in each group. Reiki or back massage were applied for 20 minutes once a day to the patients in the Reiki and back massage groups.

DETAILED DESCRIPTION:
The study was carried out to determine the effect of Reiki and back massage application on pain, analgesic use and vital signs in women underwent open abdominal hysterectomy. This study used an experimental pretest and posttest design with two experimental groups (Reiki and back massage), and a control group. The population of the study consisted of women who underwent abdominal hysterectomy in the Obstetrics Clinics of the Gazi Training and Research Hospital and Dicle University Hospital between July 2017 and February 2018. Open abdominal hysterectomy is usually performed in clinics on a planned basis.The data were collected by the researcher in the clinic by the face-to-face interview method using the Patient Information Form, the Numeric Pain Rating Scale (NPRS), and the Vital Signs and Postoperative Analgesic Follow-up Form.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery in elective conditions,
* were hospitalized for at least two days after surgery,
* did not develop any serious complications after surgery,
* were operated on under general anesthesia,
* had no previous Reiki or back massage,
* had a pain level of 3 or above according to the Numeric Pain Rating Scale,
* had no cognitive, affective or communication problems,
* used only one type of analgesic (a non-narcotic analgesic)
* did not use patient-controlled analgesics.

Exclusion Criteria:

* Patients with chronic disease (such as hypertension, cardiovascular disease),
* severe complications after surgery (such as bleeding, infection),
* those who were taking narcotic analgesics.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Open abdominal hysterectomy is usually performed in clinics on a planned basis. Patients undergoing open abdominal hysterectomy are hospitalized over 1-2 days before the surgery and they are discharged on the postoperative 3 rd day if there is no postoperative complication. Routine analgesics and antibiotics are given to all patients in the postoperative period.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-07-09 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 1st postoperative days
  This scale gives pain a numeric score, from the absence of pain (0 integers) to unbearable pain (10 integers).
Vital Signs and Postoperative Analgesic Follow-up Form (VSPAFF) | 1st postoperative days
  This consists of questions about the application of reiki and back massage, information about the patients' vital signs, including pulse rate (min), respiratory rate (min), blood pressure (mmHg) at the time of measurement, as well as information about the number and doses (milligrams) of analgesics taken postoperatively.
Numeric Pain Rating Scale (NPRS) | 2 nd postoperative days
  This scale gives pain a numeric score, from the absence of pain (0 integers) to unbearable pain (10 integers).
Vital Signs and Postoperative Analgesic Follow-up Form (VSPAFF) | 2 nd postoperative days
  This consists of questions about the application of reiki and back massage, information about the patients' vital signs, including pulse rate (min), respiratory rate (min), blood pressure (mmHg) at the time of measurement, as well as information about the number and doses (milligrams) of analgesics taken postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Hediye Utli, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
After the article is accepted for publication, it will be shared with other researchers.